CLINICAL TRIAL: NCT03065699
Title: A Multi-centre, Randomised Controlled Study, to Evaluate the Safety and Performance of The DIALIVE Liver Dialysis Device (LDD) in Patients With Acute on Chronic Liver Failure (ACLF) Versus Standard of Care (SOC)
Brief Title: Safety and Performance Trial of DIALIVE Liver Dialysis Device in Acute On Chronic Liver Failure Patients
Acronym: DIALIVE _ACLF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yaqrit Ltd (Industry)
Collaborators: European Foundation for Chronic Liver Failure (Unknown); University College, London (Other); Fakkel bvba (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: YAQ-002; CIV-16-08-016644 (Other: EUDAMED number issued by MHRA)
Record Dates: First submitted 2017-01-18; First posted 2017-02-28 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Acute on Chronic Liver Failure
Keywords: Medical device; Liver dialysis; Haemofilter; ACLF
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Intervention Model Description: The design is a multi-centre, randomised, controlled, study to generate data for the evaluation of safety (as measured by the percentage of subjects who experience at least one serious adverse event (SAE)) and performance (as measured by lowering of the plasma endotoxin concentrations, and improved albumin function) of DIALIVE in 24 evaluable patients with Acute on Chronic Liver Failure (ACLF) versus standard of care (SOC). During the study the sample size was increased to include a total 30 evaluable patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): For patients with ACLF grade 1 or 2 and randomised to the 'Standard of care' arm, the location of treatment (ICU or general ward) will be determined by their clinical need and will be decided by the site Principal Investigator. They will receive standard of care.
- DIALIVE Liver Dialysis Device treatment arm (Active Comparator): Patients with ACLF grade 1 and ACLF grade 2 on the background of alcoholic cirrhosis randomized to the DIALIVE arm will receive treatment in an intensive care (ICU) or renal dialysis unit setting. They will receive DIALIVE treatment according to a fixed treatment schedule over a period of 10 days post-randomization.
  Interventions: Device: DIALIVE Liver Dialysis Device

INTERVENTIONS:
Device: DIALIVE Liver Dialysis Device — ACLF patients will receive dialysis treatment for 8-12 hrs/day and on three to five consecutive days over a 10-day time period. Dialysis treatment is performed by using the DIALIVE device provided by YAQRIT Ltd.
  Other Names: YAQ 002
  Arms: DIALIVE Liver Dialysis Device treatment arm

SUMMARY:
The First-In-Man study is a multi-centre, randomised, controlled, study to generate data for the evaluation of safety and performance of DIALIVE Liver Dialysis Device in 24 evaluable patients with Acute on Chronic Liver Failure (ACLF) versus standard of care (SOC).

DETAILED DESCRIPTION:
The First-In-Man study will evaluate the safety and performance of DIALIVE Liver Dialysis Device in Acute on Chronic Liver Failure (ACLF) patients and will compare the outcome with patients treated under standard of care (SOC).

The hypothesis is that DIALIVE will significantly improve the prognosis of ACLF patients by modulating systemic inflammation.

The target patient population are men and women ≥18 years, ≤81yr. Patients with ACLF grade 1 and ACLF grade 2 on the background of alcoholic cirrhosis. During the study, inclusion criteria were expanded to include also AKI-1 and ACLF 3a patients. Treatment will be undertaken in an intensive care (ICU) or renal dialysis unit setting if the patients are randomised to the DIALIVE treatment arm. For patients randomised to the 'Standard of care' arm, the location of treatment (ICU or general ward) will be determined by their clinical need and will be decided by the site Principal Investigator.

This project has received funding from the European Union's Horizon 2020 research and innovation programme under grant agreement No 733057.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥18 years ≤81yr who have given informed consent to participate in the study and are able to understand and comply with the requirements of the study (otherwise written informed consent must be obtained on behalf of the subject in accordance with local ethical and legal requirements).
* History indicative of alcohol-related cirrhosis based on clinical, radiological and/or histological evidence.
* History of an acute decompensating event (including but not limited to ascites, gastrointestinal bleeding, hepatic encephalopathy and/or acute bacterial infections), occurring within ≤6 weeks of screening.
* • Subject with :

  * ACLF Grade 1, 2 or 3a defined per the CLIF-C OF scoring system OR
  * single hepatic organ failure for serum bilirubin > 20 mg/dL (342 µmol/L) at screening and randomization, OR
  * AKI-stage 1b (sCr > 1.5 mg/dL or 134 µmol/L).
* Where a subject has received corticosteroids for alcohol-induced ACLF, is unresponsive to at least 7 days of treatment (where lack of response defined as Lille score > 0.45 or steroids stopped before 7 days due to any complication such as infection). This refers to the first course of corticosteroid therapy only.

Exclusion Criteria:

* Co-infection with HIV and AIDS defining illness.
* Subjects with acute or sub-acute liver failure without underlying cirrhosis.
* Subjects with severe thrombocytopaenia, defined by the platelet count of < 40,000 / mm3 or rapid reduction in platelet count (> 50% reduction) 24 hrs prior to inclusion.
* Subjects with International Normalised Ratio (INR) > 3
* ACLF 3b patients, i.e. ACLF with more than 3 organ failures.
* Subjects with cirrhosis who develop decompensation at any time in the post-operative period following partial partial liver resection or major non-liver surgery.
* Subjects with uncontrolled infection. Patients may be entered into the study provided antimicrobials have been administered for at least 48 hours with an appropriate response observed prior to randomization.
* Subjects with respiratory organ failure (as per CLIF-C OF scoring: PaO2/FiO2< 200 mmHg or 27 kPa or SaO2/FiO2 < 214).
* Subjects with haemodynamic instability:

  i) persistent hypotension (mean arterial pressure < 65 mmHg) with evidence of tissue hypoperfusion, not responsive to volume resuscitation and/or low dose vasopressor support; ii) a norepinephrine dose of > 0.2 µg/kg/min, or a second pressor (terlipressin for variceal haemorrhage and/or hepato-renal syndrome does not count as pressor, unless it is specifically used to treat systemic hypotension) at screening or randomization. Patients can be reconsidered for study inclusion after at least a 24 hour period of norepinephrine requirement < 0.2 µg/kg/min.
* Subjects not considered appropriate for full active treatment including organ support or those with a Do Not Attempt Cardio-Pulmonary Resuscitation order (DNACPR).
* Subjects with active, or with a history of non hepatic malignancy unless adequately treated or in complete remission for five or more years.
* Patients with HCC outside Milan criteria.
* Significant systemic or major illness other than liver disease, including coronary artery disease, cerebrovascular disease, pulmonary disease, renal failure, serious psychiatric disease, that, in the opinion of the Investigator would preclude the subject from participating in and completing the study.
* Subject who has received any investigational drug or device within 30 days of dosing or who is scheduled to receive another investigational drug or device in the course of the study; concomitant observational studies are allowed.
* Evidence of uncontrolled seizures.
* Subjects diagnosed with Creutzfeldt-Jakob disease.
* In females: known pregnancy or lactating.
* Subjects weighing less than 30 kg (as per contra-indications of oXiris and septeX)
* Where subjectspresent with a known allergy to heparine of have type II thrombocytopaenia caused by heparin (HIT syndrome type II)
* In the opinion of the investigator, it is unsafe for the patient to be considered for the study.

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-07-09 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Safety of DIALIVE in terms of percentage of ACLF patients experiencing serious adverse events during DIALIVE treatment period. | Treatment period is from 1 to 10 days post-randomization.
  To evaluate the safety of the DIALIVE device in patients with Acute on Chronic Liver Failure Grades 1 and 2 (ACLF). Outcome measure is: The percentage of subjects who experience at least one (1) serious adverse event (SAE) between Day 1 and Day 10.(DIALIVE arm only).
  Outcome is measured on day 10 and compared between treatment arms.
Safety of DIALIVE in terms of percentage of ACLF patients who discontinued treatment due to severe adverse event. | Treatment period is from 1 to 10 days post-randomization.
  The outcome measure is the percentage of subjects who discontinued DIALIVE treatment due to a serious adverse device event (SADE) between Day 1 (first day of treatment) and Day 10.(DIALIVE arm only)

SECONDARY OUTCOMES:
Performance of DIALIVE by assessing removal of endotoxins. | End of DIALIVE treatment (max 10 days after randomization)
  To evaluate the performance of the DIALIVE device in patients with ACLF (DIALIVE arm only). Outcome measure is :
  - Change in Plasma endotoxin concentrations between end of treatment with DIALIVE and the beginning of treatment with DIALIVE (Day 1).
  TV: 40% reduction; AV: 20% reduction
Performance of DIALIVE by assessing removal of albumin. | End of DIALIVE treatment (max 10 days after randomization)
  To evaluate the performance of the DIALIVE device in patients with ACLF (DIALIVE arm only). Outcome measure is :
  - Change in Albumin function (Human non-mercapt albumin -2 (HNA-2) / Human mercapt albumin (HMA ratio) between end of treatment with DIALIVE and the beginning of treatment with DIALIVE (Day 1)
Change in Clinical Parameters by DIALIVE treatment (ACLF grade and score) between treatment arms. | Treatment period is from 1 to 10 days post-randomization
  Evaluate the improvement in clinical parameters between Acute on Chronic Liver Failure (ACLF) patients receiving DIALIVE treatment vs Standard of Care. Outcome measure is:
  - Change in CLIF-C score (Chronic LIver Failure Consortium)
Change in Clinical Parameters by DIALIVE treatment (ACLF grade) between treatment arms. | Treatment period is from 1 to 10 days post-randomization
  Evaluate the improvement in clinical parameters between Acute on Chronic Liver Failure (ACLF) patients receiving DIALIVE treatment vs Standard of Care. Outcome measure is:
  - Change in ACLF Grade
Change in mortality between treatment arms. | At day 28 post-randomization (for all patients). At day 90 for those patients enrolled under protocol version 6.0.
  The outcome measure is the difference in mortality between the DIALIVE treatment arm and the Standard of Care arm at day 28 post-randomization.
  During the study, the follow up period was prolonged to 90 days (3 months).
Change in Clinical Parameters by DIALIVE treatment (CLIF-C score) between treatment arms. | Treatment period is from 1 to 10 days post-randomization
  Evaluate the improvement in clinical parameters between Acute on Chronic Liver Failure (ACLF) patients receiving DIALIVE treatment vs Standard of Care. Outcome measure is:
  - Change in CLIF-C score (Chronic LIver Failure Consortium)
Status of ICU and hospital discharge. | Treatment period is from 1 to 90 days post-randomization.
  Location of patient at day 28 and 90 post randomization, and timing of discharge from hospital.
Length of stay in ICU and in hospital | Assessment is done on day 28 and day 90.
  Evaluation of length of stay of patient in the hospital and on the ICU.
ICU and hospital re-adminssions with another episode of ACLF | Assessment is done on day 28 and day 90.
  Assessment of re-admissions of patients for another episode of ACLF after hospital discharge post-randomization.

OTHER OUTCOMES:
Efficacy of the DIALIVE for liver function: changes in MELD score | Treatment period is from 1 to 10 days post-randomization
  Outcome measure as compared between SoC and DIALIVE arm is:
  * Liver: Changes in MELD score, plasma/serum cCK18/M30 and flCK18/M65 (markers of liver cell death).
  * Liver: serum bilirubine Model for End-Stage Liver Disease (MELD) Scoring Systems.
Efficacy of the DIALIVE for kidney function: changes in creatine and NGAL | Treatment period is from 1 to 10 days post-randomization
  Outcome measure as compared between SoC and DIALIVE arm is:
  - Kidney: Changes in serum creatinine and urinary NGAL (Neutrophil gelatinase-associated lipocalin - marker of kidney injury).
Efficacy of the DIALIVE for brain function: changes in West Haven Criteria | Treatment period is from 1 to 10 days post-randomization
  Outcome measure as compared between SoC and DIALIVE arm is:
  - Brain: West Haven Criteria to assess changes in severity of hepatic encephalopathy.
Efficacy of the DIALIVE for immune function. | Treatment period is from 1 to 10 days post-randomization
  Outcome measure as compared between SoC and DIALIVE arm is:
  - Immune function: Incidence of Infection. Changes in white cell count and plasma-induced neutrophil function (Phagoburst and Phagotest), serum CRP and cytokines (TNF-α, IL-6, IL-8, IL-10, IL1RA).
Assessment of coagulation and haemostasis. | Treatment period is from 1 to 10 days post-randomization
  Outcome measure as compared between SoC and DIALIVE arm is:
  - Coagulation: Changes in INR and platelet levels.
Efficacy of the DIALIVE for pulmonary function. | Treatment period is from 1 to 10 days post-randomization
  Outcome measure as compared between SoC and DIALIVE arm is:
  - Lung: P/F or S/F ratio.
Efficacy of the DIALIVE for the cardiovascular function. | Treatment period is from 1 to 10 days post-randomization
  Outcome measure as compared between SoC and DIALIVE arm is:
  - Cardiovascular system: measurement off the Mean Arterial Pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Banwari Agarwal, Dr, Principal Investigator — Royal Free Hospital London NHS
Locations (12):
- university Hospital Graz, Graz, Austria
- University Hospital Erasmus, Brussels, Belgium
- University Hospital, Aarhus, Denmark
- France (2):
  - Hôpital Beaujon, Clichy
  - Paul Brousse Hospital, Villejuif
- University Hospital of Rostock, Rostock, Germany
- Fundeni Clinical Institute, Bucharest, Romania
- Spain (2):
  - Hospital Clinic Barcelona, Barcelona
  - University Hospital Gregorio Maragnon, Madrid
- United Kingdom (3):
  - Royal Free Hospital London NHS, London, Hampstead
  - university hospital BASILDON, Basildon
  - Queens Medical Centre, Nottingham

IPD SHARING:
Plan to Share IPD: No
Only anonymized clinical data can be shared out of central database according to the H2020 project plan.

REFERENCES:
- [Background] Lee KC, Baker LA, Stanzani G, Alibhai H, Chang YM, Jimenez Palacios C, Leckie PJ, Giordano P, Priestnall SL, Antoine DJ, Jenkins RE, Goldring CE, Park BK, Andreola F, Agarwal B, Mookerjee RP, Davies NA, Jalan R. Extracorporeal liver assist device to exchange albumin and remove endotoxin in acute liver failure: Results of a pivotal pre-clinical study. J Hepatol. 2015 Sep;63(3):634-42. doi: 10.1016/j.jhep.2015.04.020. Epub 2015 May 1. PMID 25937432
- [Derived] Agarwal B, Canizares RB, Saliba F, Ballester MP, Tomescu DR, Martin D, Stadlbauer V, Wright G, Sheikh M, Morgan C, Alzola C, Lavin P, Green D, Kumar R, Sacleux SC, Schilcher G, Koball S, Tudor A, Minten J, Domenech G, Aragones JJ, Oettl K, Paar M, Waterstradt K, Bode-Boger SM, Ibanez-Samaniego L, Gander A, Ramos C, Chivu A, Stange J, Lamprecht G, Sanchez M, Mookerjee RP, Davenport A, Davies N, Pavesi M, Andreola F, Albillos A, Cordingley J, Schmidt H, Carbonell-Asins JA, Arroyo V, Fernandez J, Mitzner S, Jalan R. Randomized, controlled clinical trial of the DIALIVE liver dialysis device versus standard of care in patients with acute-on- chronic liver failure. J Hepatol. 2023 Jul;79(1):79-92. doi: 10.1016/j.jhep.2023.03.013. Epub 2023 May 31. PMID 37268222
- See also: webpage legal responsible partner & spnosor — http://yaqrit.com
- Available data/document: Clinical Study Report: DIALIVE CSR summary 20210319 — http://yaqrit.com — A summary of the final Clinical Study Report can be obtained through request to: 1. YAQRIT Ltd, attention of Daniel Green, CEO (daniel.green@yaqrit.com) or Carrie Morgan (carrie.morgan@yaqrit.com) 2. FAKKEL bvba, attention of Jaak Minten, CEO (info@fakkel-bvba.com)

DOCUMENTS (3):
  • Study Protocol (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT03065699/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/99/NCT03065699/SAP_001.pdf
  • Informed Consent Form (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT03065699/ICF_002.pdf